CLINICAL TRIAL: NCT07003763
Title: The Effect and Safety of Electroacupuncture on Treating Cancer-related Depression: a Randomized Controlled Clinical Trial
Brief Title: Electroacupuncture on Treating Cancer-related Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acupuncture Dep
Record Dates: First submitted 2025-05-14; First posted 2025-06-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Depression; Cancer
Keywords: Electroacupuncture; cancer; depression; randomized controlled trial
MeSH Terms: conditions — Depression; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Active Comparator): Participants in the electroacupuncture group will receive treatment based on a semi-standardized acupuncture protocol, which includes six main acupoints and two supplementary acupoints selected based on individual symptom presentation.
  Interventions: Device: Electroacupuncture treatment; Other: Standard care
- sham acupuncture group (Placebo Comparator): Participants in the control group will receive superficial acupuncture at non-acupoint, non-meridian locations as placebo control.
  Interventions: Other: Superficial acupuncture at Non-Acupoints; Other: Standard care

INTERVENTIONS:
Device: Electroacupuncture treatment — Participants in this group will receive electroacupuncture (EA) based on a semi-standardized protocol. Each treatment session will involve needling at six main acupoints and two supplementary points, selected based on individual symptoms.
  * Main acupoints: Baihui (GV20), Yintang (EX-HN3), Guanyuan (CV4), Qihai (CV6), bilateral Zusanli (ST36), bilateral Sanyinjiao (SP6).
  * Supplementary acupoints: Selected from Shenting (GV24), Sishencong (EX-HN1), Fengchi (GB20), Neiguan (PC6), Hegu (LI4), Shenmen (HT7), Yanglingquan (GB34), Taixi (KI3), and Taichong (LR3).
  All patients will be placed in the supine position. After routine disinfection of all acupoints using 75% alcohol, needles will be inserted using a gentle tapping technique. Once Deqi sensation is achieved, three pairs of electrodes from an EA device will be connected to the handles of the needles at Baihui and Yintang, and bilaterally at Zusanli and Sanyinjiao. Each treatment session will last for 30 minutes.
  Arms: Electroacupuncture group
Other: Superficial acupuncture at Non-Acupoints — Participants in this group will receive superficial acupuncture at six pseudo-acupoints that do not correspond to any recognized meridian or traditional acupoint. These points are anatomically matched in location (head, upper limbs, lower limbs, and trunk) to the main acupoints used in the EA group but are located at non-meridian, non-acupoint sites in a horizontal position. Acupuncture needles will be connected to an electroacupuncture device with broken wires and thus no electrical stimulation is actually delivered.
  All patients will be placed in a supine position. After routine disinfection of the selected sites using 75% alcohol, sterile disposable filiform needles (0.22 × 25 mm) will be lightly inserted to a depth of approximately 3 mm without requiring deqi. The needles will be applied using a gentle tapping technique at non-meridian, non-acupoint locations. The needle will be retained for 30 minutes. The session frequency and total treatment course will match the EA group.
  Arms: sham acupuncture group
Other: Standard care — All participants, regardless of group assignment, will receive standard care as part of routine oncological and psychological management. Standard care includes:
  * Basic psychological support: General psychological counseling or emotional support provided by nursing staff or clinical psychologists as needed, without structured psychotherapy or pharmacological antidepressant interventions unless clinically indicated.
  * Health education: Guidance on sleep hygiene, nutrition, and stress management, along with education about cancer-related emotional symptoms and coping strategies.
  * Medication management: Participants will continue their current medications for chronic comorbidities (e.g., antihypertensives, antidiabetics) as previously prescribed. However, cancer-related medications associated with active treatment-such as chemotherapy, targeted therapies, immunotherapy, or hormonal therapy-will be excluded during the trial period to avoid confounding effects.

SUMMARY:
Cancer-related depression (CRD) is a common psychological condition among cancer patients during diagnosis, treatment, and recovery, and is associated with reduced quality of life, impaired immune function, and poorer clinical outcomes. As cancer incidence and mortality continue to rise in China, the psychological burden on patients is receiving increasing attention. Electroacupuncture (EA) has shown potential in treating various types of depression and related somatic symptoms, but evidence regarding its efficacy, safety, and long-term effects in CRD remains limited. This randomized controlled trial aims to evaluate the short- and long-term efficacy and safety of EA for CRD, with the goal of providing evidence to support effective and optimized treatment strategies.

DETAILED DESCRIPTION:
Cancer-related depression (CRD) is a prevalent and complex comorbidity among cancer patients, often arising during diagnosis, treatment, or disease progression. It is associated with a range of psychological and somatic symptoms that significantly reduce quality of life, compromise treatment adherence, and may negatively affect clinical outcomes and overall survival. As cancer incidence and mortality continue to rise in China's aging population, addressing the emotional and psychological burden of cancer has become increasingly important.

Current treatments for CRD largely rely on pharmacological interventions, particularly selective serotonin reuptake inhibitors (SSRIs). However, these medications often have delayed onset, potential side effects, and limited tolerability in patients undergoing cancer treatment. These limitations highlight the need for safe, non-pharmacological alternatives that can effectively alleviate depressive symptoms in this vulnerable population.

Acupuncture, a traditional Chinese medical therapy, has been widely used for managing depressive disorders and cancer-related symptoms. Electroacupuncture (EA), which combines needling with electrical stimulation, has demonstrated therapeutic potential in preliminary studies for depression and symptom relief in cancer patients. Despite encouraging results, the overall quality of evidence remains low, and rigorous randomized controlled trials (RCTs) focusing specifically on CRD are still lacking.

This study aims to evaluate the efficacy and safety of electroacupuncture in the treatment of CRD through a well-designed, randomized, assessor-blinded controlled trial. The trial will assess both short-term and long-term outcomes in patients with clinically diagnosed CRD, using validated measures for depression severity, quality of life, and symptom burden. Participants will be randomly assigned to either an intervention or control group, and all participants will continue to receive routine care during the study.

The results of this trial will contribute to the growing body of evidence on integrative approaches in cancer care. It aims to determine whether EA can serve as a safe and effective adjunct to conventional cancer treatment, improve patients' emotional well-being, and support a more holistic model of care. This research also aligns with national health strategies promoting integrative medicine and may inform future clinical guidelines for managing psychological distress in cancer populations.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of depression attributed to cancer itself or cancer-related treatments, meeting the diagnostic criteria for depressive disorder（DSM-V).
2. Age between 18 and 75 years, regardless of sex.
3. Hamilton Depression Rating Scale-17 (HDRS-17) total score >17 at baseline.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2.
5. No previous exposure to acupuncture treatment.
6. Ability to understand the study procedures and willingness to provide written informed consent.

Exclusion Criteria:

1. Planned to undergo surgery, chemotherapy, radiotherapy, immunotherapy, or other active cancer-related treatments during the study period.
2. History of major depressive episodes prior to cancer diagnosis.
3. Pain Rating Index (PRI) score ≥4 due to cancer-related pain.
4. Estimated life expectancy of 12 months or less.
5. Presence of severe ulcers, abscesses, or active skin infections at or near the acupuncture sites.
6. Clinically significant dysfunction of major organs, including severe cardiac, cerebral, hepatic, renal impairment; decompensated pulmonary disease; or other serious systemic illnesses.
7. Pregnant or breastfeeding women.
8. Participation in another clinical trial within the past 30 days.
9. Patients with a cardiac pacemaker or other implanted electronic medical devices.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale - 17 items | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24.
  The HDRS-17 is a clinician-administered scale widely used to assess the severity of depressive symptoms and evaluate treatment efficacy in clinical trials. In this study, the HDRS-17 will be administered by trained raters using structured clinical interviews. The total score ranges from 0 to 52, with higher scores indicating more severe depression. A total score >17 is considered to reflect at least moderate depression, while a score ≤7 is typically interpreted as remission. Higher scores represent greater symptom severity.

SECONDARY OUTCOMES:
Remission Rate | Week 12
  Proportion of participants with Hamilton Depression Rating Scale - 17 items score <8 at Week 12.
Response Rate | Week 12
  Proportion of participants with ≥50% reduction from baseline in Hamilton Depression Rating Scale - 17 items score at Week 12.
Patient Health Questionnaire-9 | Baseline, Week 12, Week 24.
  The PHQ-9 is a self-administered instrument used to screen for depression severity and monitor treatment response. It consists of 9 items, each corresponding to DSM-5 criteria for major depressive disorder, rated on a 4-point Likert scale (0 = "not at all" to 3 = "nearly every day"). The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms. Score interpretation is as follows: 5-9 = mild, 10-14 = moderate, 15-19 = moderately severe, and 20-27 = severe depression. A reduction in score over time will be used to assess treatment efficacy.
Pain Rating Index | Baseline, Week 12, and Week 24.
  The Pain Rating Index (PRI) is derived from the Short-Form McGill Pain Questionnaire (SF-MPQ) and is used to evaluate the intensity and quality of pain. It includes 15 descriptors (11 sensory and 4 affective), each rated on a 4-point scale: 0 = "none", 1 = "mild", 2 = "moderate", and 3 = "severe". The PRI is calculated by summing the scores of the individual descriptors, providing a composite measure of both sensory and affective pain dimensions. A higher PRI score indicates more severe pain experience.
Quality of Life Questionnaire for Cancer Patients | Baseline, Week 12, and Week 24.
  The EORTC QLQ-C30 is a validated, cancer-specific instrument designed to assess health-related quality of life in oncology patients. It comprises five functional scales (physical, emotional, social, cognitive, and role functioning), a global health status/quality of life scale, three symptom scales (fatigue, nausea/vomiting, and pain), and several single items assessing additional symptoms (e.g., dyspnea, appetite loss, insomnia, constipation, diarrhea) and financial impact. Each item is rated using a 4-point Likert scale (1 = "not at all" to 4 = "very much"), except for the global health scale, which uses a 7-point numeric scale. Scores are linearly transformed to a 0-100 scale. Higher scores on functional and global health scales indicate better functioning and quality of life, while higher scores on symptom scales represent greater symptom burden.
Use of Antidepressants | Baseline, and Week 12.
  Documented dosage and frequency of antidepressant medication usage through patient-reported medication diaries.
Treatment Emergent Symptom Scale (TESS) | Through study completion, an average of 6 months
  The Treatment Emergent Symptom Scale (TESS) is a clinician-rated tool used to systematically evaluate adverse events and treatment-emergent side effects during the course of clinical trials. Symptoms are rated based on presence, severity, and clinical relevance. Each item is scored to reflect the degree of discomfort and interference with function.

CONTACTS AND LOCATIONS:
Overall Officials: Shifen Xu, Doctor, Study Director — SHMTCM's Acupuncture Department
Locations (1):
- Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No